CLINICAL TRIAL: NCT02002676
Title: Prevalence and Outcome of Hypermetabolism in Initial Phase of Intensive Care Unit Patient: a Prospective Observational Study
Brief Title: Prevalence and Outcome of Hypermetabolism in Initial Prevalence and Outcome of Hypermetabolism in Initial Phase of Intensive Care Unit Patient: a Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing University School of Medicine (Other)
Collaborators: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Chao Wu, Ph.D.candidate, Nanjing University School of Medicine
Other Study IDs: 2013KLY-022
Record Dates: First submitted 2013-11-26; First posted 2013-12-06 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: SIRS; Sepsis; Septic Shock
Keywords: rest energy expenditure,critical ill, outcome
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients in critical illness frequently present hypermetabolism， which can extremely increase the rest energy expenditure（REE）. We hypothesize that if we alleviate the extremely increased REE will improve ICU patients' outcome

DETAILED DESCRIPTION:
This study focuses on the early changes of REE of critical ill patients when they admitted to ICU.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 year.
* APACHEⅡ score≥8

Exclusion Criteria:

* Hypercortisolism
* Thyroid disease
* Tracheoesophageal fistula
* FiO2>60 or PEEP>12cm H2O in mechanical ventilate
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who admitted ICU with hypermatebolic status, which the results of indirect calorimetry show that the actual rest energy expenditure values are remarkably higher than the predicted ones.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Mortality rate of 28 days | From ICU admission to 28th days of observation

SECONDARY OUTCOMES:
Incidence of Multiple Organ Dysfunction Syndrome（MODS）in 60 days | From ICU admission to 60th days of observation

OTHER OUTCOMES:
Length of stay in ICU | Length of ICU stay within 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Wang, MD, Study Director — Nanjing University School of Medicine
Locations (1):
- Nanjing University School of Medicine, Nanjing, Jiangsu, China